CLINICAL TRIAL: NCT00793247
Title: A Double-Blind, Placebo-Controlled, Cross-Over, Multiple (n=1) Trial to Evaluate the Effects of R093877 in Patients With Chronic Intestinal Pseudo-Obstruction (CIP).
Brief Title: Efficacy Study of Prucalopride to Treat Chronic Intestinal Pseudo-Obstruction (CIP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Movetis (Industry)
Other Study IDs: GBR-7
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Intestinal Pseudo-Obstruction

INTERVENTIONS:
Drug: PRU-PLA-PRU-PLA
Drug: PLA-PRU-PLA-PRU
Drug: PLA-PRU-PRU-PLA
Drug: PRU-PLA-PLA-PRU

SUMMARY:
This study was designed to investigate the clinical safety, tolerability and efficacy of prucalopride in improving the symptoms associated with chronic intestinal pseudo-obstruction (CIP) in subjects with CIP. The study hypothesis was that prucalopride at doses up to 4 mg is safe, well tolerated, efficacious and improves the symptoms associated with CIP.

DETAILED DESCRIPTION:
This phase II, double-blind, placebo-controlled, two-treatment four periods cross-over trial investigated the clinical safety, tolerability and the efficacy of R093877 (prucalopride) in improving the symptoms associated with chronic intestinal pseudo-obstruction (CIP) in subjects with CIP.

Subjects were treated for 4 periods of 12 weeks each with either R093877 2 mg (2 periods) or placebo (2 periods). In each of the first and second 6 month period, there was a placebo (PLA) and an active drug (PRU) treatment period. There were no wash-out periods. In total,7 subjects were randomized; 2 were assigned to the PLA-PRU-PLA-PRU, 2 to the PRUPLA-PRU-PLA, 2 to the PLA-PRU-PRU-PLA, and 1 to the PRU-PLA-PLA-PRU sequence group. Subjects were allowed to use up to 4 mg of prucalopride per day if the 2 mg dose seemed to be insufficient. Two subjects used an average of 3 mg of prucalopride per day during the active drug periods.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years;
* A history of chronic pseudo-obstruction for at least 3 months;
* Subjects with chronic idiopathic pseudo-obstruction or chronic pseudo-obstruction secondary to scleroderma or intestinal polyneuropathy;
* CIP had been diagnosed by a Barium-imaging study showing the presence of dilatation of any part of the small bowel (with or without the presence of large bowel dilatation);

Exclusion Criteria:

* Subjects with organic obstructing lesions causing intestinal obstruction;
* Current uncontrolled cardiovascular or lung disease, neurologic or psychiatric disorders (including substance abuse but with the exception of nicotin), alcoholism, cancer or AIDS and endocrine disorder;
* Impaired renal function
* A serum amylase, a serum glutamic-oxaloacetic transaminase (SGOT) or a serum glutamic-pyruvic transaminase (SGPT)concentration of > 2 times the normal limit;
* Laboratory values outside the reference range of the laboratory, unless explained by the disease or felt by the investigator to be clinically unimportant;
* Use of disallowed concomitant therapy;
* Female subjects who were pregnant or wished to become pregnant during the course of the trial or who were lactating;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Northwick Park Hospital, London, United Kingdom